CLINICAL TRIAL: NCT07093879
Title: EFFECT OF STATIC HAMSTRING STRETCHING ON DYNAMIC BALANCE, FOOT POSTURE AND FUNCTION IN INDIVIDUALS WITH PRONATED FEET
Brief Title: Hamsrting Stretching on Dynamic Balance, Foot Posture and Function in Pronated Feet.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Donia Mohamed Abd Elfattah Sanad, demonstrator at faculty of physical therapy kfs university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005455
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pronation; Ankle
Keywords: Pronated Foot, DYNAMIC BALANCE, STATIC HAMSTRING STRETCHING

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): 14 individuals will receive static hamstring stretching three treatment sessions per a week, short foot exercise (SFE), towel curl exercise (TCE), toe spread-out exercise (TSO) daily, tibialis posterior strengthening, gluteal muscles strengthening 3 times per week for 6 weeks.
  Interventions: Other: STATIC HAMSTRING STRETCH
- GROUP B (Other): 14 individuals will receive SFE, TCE, TSO daily, tibialis posterior strengthening, gluteal muscles strengthening 3 times per week for 6 weeks.
  Interventions: Other: STATIC HAMSTRING STRETCH

INTERVENTIONS:
Other: STATIC HAMSTRING STRETCH — For the static stretching technique, individuals lay supine in a straight posture on the treatment table and relaxed. Then, the pelvis and thighs opposite to the lower limb to which the stretching technique was to be applied were tied with Velcro straps. With the knees extended, the foot in neutral position and the hip joint bent as much as possible within its range, the hip joints were bent more until the hamstring muscle was stretched with light, tolerable pain, and kept there for 30 seconds

SUMMARY:
Foot pronation is a natural and essential movement that occurs during walking or running. It involves the inward rolling of the foot, allowing for effective shock absorption and weight distribution, Individuals with pronated feet have poorer standing postural control compared with individuals with normal feet. This may be due to the reduced stability within the foot joints. Static stretching (SS) has been shown to increase the joint ROM, improve performance, and prevent injury. The connection between the hamstring muscles and the intrinsic foot muscles is explained through their integration within the same myofascial pathway-the superficial back line.

DETAILED DESCRIPTION:
Over-pronated foot is responsible for up to 60-90% of all foot and lower extremity pathologies associated with overuse injuries. This biomechanically abnormal foot posture alters the normal transitions of the subtalar joint required during dynamic activities. Therefore, deviations of the foot from its normal posture, place the foot under excessive stress and demand on the postural control .

The hamstring muscles, as the primary flexors of the knee, play a crucial role in maintaining balance due to their involvement across both the hip and knee joints. Limited flexibility in this muscle group can negatively impact balance performance and increase the risk of lower extremity injuries, pelvic and spinal misalignment, hip immobility, and pain. Stretching is a commonly used method to enhance joint range of motion and muscle extensibility, which supports injury prevention and rehabilitation, and may also improve balance through various physiological mechanisms .

Static hamstring stretching may lead to improved gait mechanics, enhanced stability, and reduced discomfort during weight-bearing activities due to the fascial connection between the hamstring muscle and plantar foot muscles, so incorporating static hamstring stretching into the physiotherapy program for individuals with pronated feet may alter foot posture, improve the dynamic balance and lower the risk of injuries associated with pronated feet.

Several techniques have been applied for improving dynamic balance and foot posture, but there was a gap in the previous literatures about using static hamstring stretch in rehabilitation of pronated feet, so this study will be conducted to determine effect of static hamstring stretch on dynamic balance and foot posture in pronated feet individuals.

ELIGIBILITY:
Inclusion Criteria:

* 1-Individual's age ranged from 18-25 years old both genders. 2- Individuals had bilateral pronated feet posture according to the navicular drop test by Brody method .

  3- individuals had bilateral hamstring tightness assessed by active knee extension (AKE) test .

  4- Body Mass Index (BMI) ranged from 18.5 to 25 kg/ m2 .

Exclusion Criteria:

- - Repeated lower extremity injuries as fractures or deformities. 2- History of surgery to the lower extremity. 3- Any neurological deficit affecting balance. 4-Any medication can affect the balance. 5- pregnant and breast feeding females. 6- fixed flat foot 7- Individuals with unilateral pronated foot. 8- Sleep disorders or chronic fatigue conditions (e.g., insomnia, chronic fatigue syndrome).

9- Uncontrolled diabetes (especially with peripheral neuropathy). 10- Visual impairments (e.g., uncorrected vision problems, glaucoma, or macular degeneration).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
DYNamic balance | 6months
  The process that maintains the center of gravity within the body's support base